CLINICAL TRIAL: NCT06880848
Title: A Prospective, Open-Label, Single-Arm, Multi-Center, Phase IV Efficacy and Safety Study of Sonidegib in Adult Patients With Locally Advanced Basal Cell Carcinoma (laBCC) in China
Brief Title: Sonidegib in Adult Patients With Locally Advanced Basal Cell Carcinoma (laBCC) in China
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jemincare (Industry)
Collaborators: Sun Pharmaceutical Industries Limited (Industry); Zhejiang Hangyu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AM20220301
Record Dates: First submitted 2025-03-12; First posted 2025-03-18 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Carcinoma, Basal Cell (BCC)
Keywords: BCC; Basal Cell Carcinoma
MeSH Terms: conditions — Carcinoma; Carcinoma, Basal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sonidegib Phosphate Capsules (Experimental): Participants will receive continuous treatment with oral administration once a day until conditions for treatment termination are met.
  Interventions: Drug: Sonidegib Phosphate Capsules

INTERVENTIONS:
Drug: Sonidegib Phosphate Capsules — Sonidegib should be taken 1 hour before or 2 hours after a breakfast

SUMMARY:
This is a Phase IV, single arm, multicenter study designed to evaluate the efficacy and safety profile of Sonidegib in chinese participants with locally advanced basal cell carcinoma (laBCC) who are not amenable to radiation therapy, curative surgery or other local therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older.
2. Patients with a histologically confirmed diagnosis of laBCC that is not amenable to radiation therapy, curative surgery, or other local therapies. Patients with laBCC must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension as ≥ 10 mm, with MRI/CT scan or on color photographs.
3. ECOG PS Score ≤ 2.
4. Patients with adequate bone marrow, liver and renal function.
5. Written informed consent obtained prior to any screening procedures.
6. Patients are willing and able to comply with the scheduled visits, treatment plan, laboratory testing, study procedures, and restrictions.
7. Females of childbearing potential agree to use contraception during treatment and for 20 months following the last dose; male patients (even after vasectomy) agree to use contraception during treatment and for 8 months after the last dose.

Exclusion Criteria:

1. Subjects in the opinion of the investigator are immunosuppressed (e.g., organ transplant recipients, HIV, systemic invasive malignancy within past 5 years excluding Stage I cervical cancer, ductal carcinoma in situ of the breast or CLL stage 0, graft vs. host disease, etc.).
2. LaBCC patients with skin lesions in multiple body locations will not be considered metastatic patients. LaBCC patients with positive (histological confirmation of BCC) regional nodal disease will be considered to have metastatic disease.
3. Poorly controlled diabetes mellitus (as per Investigator's discretion in consultation with Sponsor's medical monitor).
4. Major surgery within 4 weeks prior to study treatment.
5. Patients with concurrent uncontrolled medical conditions that may interfere with their participation in the study or potentially affect the interpretation of the study data.
6. Patients unable to take oral drugs or with lack of physical integrity of the upper gastrointestinal tract or known malabsorption syndromes.
7. Patients who have previously been treated with systemic Sonidegib or with other Hh pathway inhibitors.
8. Patients who have neuromuscular disorders (e.g. inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis and spinal muscular atrophy).
9. Patients who are planning on embarking on a new strenuous exercise regimen after initiation of study treatment.
10. Have participated in other clinical trials within 4 weeks prior to the first dose of sonidegib.
11. Have received other anti-neoplastic therapy within 4 weeks prior to study treatment.
12. Patients who are receiving medications known to be moderate and strong inhibitors or inducers of cytochrome P450 (CYP) 3A4/5 or drugs metabolized by CYP2B6 or CYP2C9 that have narrow therapeutic index, and that cannot be discontinued before starting treatment with sonidegib. Medications that are strong CYP3A4/5 inhibitors should be discontinued at least 7 days and strong CYP3A/5 inducers for at least 2 weeks prior to starting treatment with sonidegib.
13. Pregnant or nursing (lactating) women, confirmed by a positive hCG laboratory test (> 5mIU/mL).
14. Unwilling or unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2023-06-21 (Actual); Primary Completion 2025-08-26 (Actual); Study Completion 2025-08-26 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | up to 1 year
  Objective response rate (ORR) is defined as the percentage of participants with a confirmed complete or partial response (CR or PR) , per modified Response Evaluation Criteria in Solid Tumors (mRECIST) as assessed by central review.

SECONDARY OUTCOMES:
Duration of Response (DoR) | up to 1 year
  The DOR for a responder is defined as the time from the participant's initial CR or PR to the first date of either disease progression or death, whichever occurs first. CR, PR and PD will be determined per mRECIST by investigator and central review, respectively
Complete response rate (CRR) per central and investigator review | up to 1 year
  CRR is defined as the percentage of participants who achieved a complete response per mRECIST
Progression-free Survival (PFS) | up to 1 year
  PFS is defined as the time from the participant's first dose of study treatment to the first date of either disease progression or death, whichever occurs first. Disease progression will be determined per mRECIST by investigator and central review, respectively
Time to tumor response (TTR) | up to 1 year
  TTR is defined as the time from the participant's first dose of study treatment to the date of initial CR or PR. CR and PR will be determined per mRECIST by investigator and central review, respectively.
Adverse event (AE)/Serious adverse event (SAE)/Treatment emergent adverse event (TEAE) | up to 1 year
  Adverse events, and changes from baseline in vital signs,etc

CONTACTS AND LOCATIONS:
Overall Officials: Hang Li, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, China, China

IPD SHARING:
Plan to Share IPD: No